CLINICAL TRIAL: NCT02014155
Title: Effects of Inspiratory Muscle Training on Respiratory Electromyographic Activity in Patients With COPD Participants and Non-participants of a Pulmonary Rehabilitation Program
Brief Title: Inspiratory Muscle Training and Respiratory Electromyographic Activity in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santa Cruz do Sul (Other)
Responsible Party: Principal Investigator, Diogo Fanfa Bordin, Scientific Initiation Scholarship, University of Santa Cruz do Sul
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UNISC_001
Record Dates: First submitted 2013-11-03; First posted 2013-12-18 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group Pulmonary Rehabilitation (Experimental): Pulmonary Rehabilitation consists of isotonic exercises of upper and lower limbs, 20-minute workout on cycle ergometer in standard desinsuflativo (expiration at the time of muscle contraction), is performed three times a week for eight weeks.
  Interventions: Other: Pulmonary Rehabilitation
- Group TMI + Pulmonary Rehabilitation (Experimental): Will be held inspiratory muscle training associated with a pulmonary rehabilitation program. The inspiratory muscle training is performed with a load of 40 to 50% of the muscle strength of the subjects. Pulmonary Rehabilitation consists of isotonic exercises of upper and lower limbs, 20-minute workout on cycle ergometer in standard deflation (expiration at the time of muscle contraction), is performed three times a week for eight weeks.
  Interventions: Other: Inspiratory Muscle Training; Other: Pulmonary Rehabilitation
- Control Group (Experimental): Inspiratory muscle training will be held three times a week for eight weeks
  Interventions: Other: Inspiratory Muscle Training
- COPD group not rehabilitation (Experimental)
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — Will be held inspiratory muscle training associated with a pulmonary rehabilitation program. The inspiratory muscle training is performed with a load of 40 to 50% of the muscle strength of the subjects.
  Arms: COPD group not rehabilitation; Control Group; Group TMI + Pulmonary Rehabilitation
Other: Pulmonary Rehabilitation — Pulmonary Rehabilitation consists of isotonic exercises of upper and lower limbs, 20-minute workout on cycle ergometer in standard deflation (expiration at the time of muscle contraction), is performed three times a week for eight weeks.
  Arms: Group Pulmonary Rehabilitation; Group TMI + Pulmonary Rehabilitation

SUMMARY:
Intended to treat disorders of the respiratory muscles can use the device Threshold IMT ® through an inspiratory muscle training (IMT) that allows training of the inspiratory muscles, the chief of these being the diaphragm which is which objectified the improvement of its function . To monitor the action of the respiratory muscles can be used several tools such as manometer that aims to assess respiratory pressures, ie, the strength of respiratory muscles, or the Surface Electromyography (sEMG) that allow evaluating the electromyographic activity of muscles analyzed. From a quantitative clinical trial, randomized and blinded, composed of 45 individuals obtained by random convenience and divided into three groups, COPD participating in a pulmonary rehabilitation program (RP) which will make TMI (TGR - Trained Group Rehabilitated), COPD does not participant in a PR program (TGNR - Trained Group not Rehabilitated) and a control group composed of healthy individuals (CG) that seek to analyze the electromyographic activity of sternocleidomastoid (SCM) and diaphragm muscle strength, lung volumes and breathing patterns before and after a period of eight weeks of TMI. Manual will also be held dynamometry to compare the grip strength of the CG, TGR and TGNR only at baseline.

Hypothesis:

1. The Inspiratory Muscle Training (IMT) increases the maximal inspiratory pressure (MIP) in COPD patients regardless of whether they are enrolled in a program of pulmonary rehabilitation (PR).
2. TMI alters the breathing pattern in COPD patients regardless of whether they were entered into a PR program.
3. Patients with COPD who do not participate in a PR program have higher handgrip strength compared to patients who did not participate in a PR program.
4. There is decreased activity of the sternocleidomastoid muscle due to increased activity in the diaphragmatic muscle fibers after a period of TMI.
5. TMI in COPD patients participating in a program RP produces greater increase in MIP, the handgrip strength, improves breathing pattern and a greater reduction in the activity of the SCM muscle and diaphragm than in those who did not participate in a program RP.
6. There will be a reduction in respiratory rate, heart rate, systolic and diastolic blood pressure and increased oxygen saturation at the end of the TMI.
7. TMI reduce the degree of dyspnea reported by patients as MRC scale at the end of the training period.

ELIGIBILITY:
Inclusion Criteria:

* Will be included in the study subjects of both sexes aged between 40 and 80 years. For the control group will participate in healthy subjects, non-smokers with normal lung function. For Group TMI + Rehabilitation, Non-Rehabilitated and Rehabilitation Group participate COPD patients with GOLD staging II and III, participants and non-participants of a PR program respectively, where individuals not participating (GTMINR) will be those who will enter the PR program during the stipulated time of study and the participants have (GTMIR) should be included in the project for at least eight weeks, the time required for a program to provide RP's effects in COPD

Exclusion Criteria:

* Not participate in the study and Group TMI + Rehabilitation, Non-Rehabilitated and Rehabilitation Group, individuals who do not fit the criteria for GOLD in stages II and III, which are in acute disease, presenting hemodynamic instability, aneurysm, cognitive impairment or any other co-morbidity that prevents this study. For the GC will not participate smokers, ex-smokers or who have compromised lung function, individuals participating in regular physical activity, ie three or more times per week, and no pathology that affects the cardiorespiratory system. Also excluded are those who do not sign the consent form.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-11-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Muscle electromyographic activity of the accessory Inspiration | The electromyographic activity will be evaluated during the inspiratory cycles for one minute, It will be evaluated over eight weeks

SECONDARY OUTCOMES:
Inspiratory Muscle Training | Will be performed with frequency of three days non-consecutive week, for eight weeks
Assessment of lung volumes | will be performed previously to the study and at the end, over eight weeks
assessment of respiratory muscle strength | will be performed previously to the study and at the end, as well as weekly to adjust the pressure load, It will be evaluated over eight weeks
breathing pattern assessment | will be performed previously to the study and at the end of the same, It will be evaluated over eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dulciane N Paiva, Doctor, Principal Investigator — University of Santa Cruz do Sul; Diogo F Bordin, Academic, Principal Investigator — University of Santa Cruz do Sul; Dannuey M Cardoso, Master, Study Director — University of Santa Cruz do Sul; Andrea LG da Silva, Doctor, Study Director — University of Santa Cruz do Sul
Locations (1):
- Universidade de Santa Cruz do Sul, Santa Cruz do Sul, Rio Grande do Sul, Brazil